CLINICAL TRIAL: NCT03347981
Title: Clinical Study to Compare Visual Performance of Two Trifocal IOLs With Different Material (Hydrophobic and Hydrophilic)
Brief Title: Clinical Study to Compare Visual Performance of Two Trifocal IOLs
Acronym: PHY1702
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beaver-Visitec International, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PHY1702
Record Dates: First submitted 2017-09-26; First posted 2017-11-20 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-05

CONDITIONS: Cataract; Lens Opacities; Presbyopia
Keywords: Intraocular Lens; trifocal; hydrophobic; hydrophilic
MeSH Terms: conditions — Cataract; Presbyopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IOL implantation experimental (Experimental): hydrophobic, trifocal intraocular lens POD F GF
  Interventions: Device: IOL implantation experimental
- IOL implantation active comparator (Active Comparator): hydrophilic, trifocal intraocular lens POD F
  Interventions: Device: IOL implantation active comparator

INTERVENTIONS:
Device: IOL implantation experimental — Implantation of trifocal IOL POD F GF consisting of hydrophobic material
  Arms: IOL implantation experimental
Device: IOL implantation active comparator — Implantation of trifocal IOL POD F consisting of hydrophilic material
  Arms: IOL implantation active comparator

SUMMARY:
Prospective, randomised, controlled, single-surgeon, single-center post-market clinical follow up study to compare the clinical outcomes of two trifocal IOLs with different material

DETAILED DESCRIPTION:
This is a prospective, randomised, controlled, single-surgeon, single-center post-market clinical follow up study whereby patients undergoing routine cataract surgery will have bilateral implantation of trifocal intraocular lenses. The patients will either be implanted with the hydrophobic IOL FineVision POD F GF or the hydrophilic IOL FineVision Pod F.

The primary and secondary effectiveness data for visual acuity, contrast sensitivity, halometry, aberrometry, questionnaire outcomes and any adverse events will be collected.

Subjects participating in the trial will attend a total of 10 study visits (1 preoperative, 2 operative and 7 postoperative) over a period of 3 months. Subjects would have the option for unscheduled visits if required medically.

Primary endpoint data will be collected at the 3 months follow up visit. Data analyses will be done after the last patient finished the final examination to support the study publication plan.

ELIGIBILITY:
Inclusion Criteria:

* Cataractous eyes with no comorbidity
* Spontaneously emitting the desire for spectacle independence after surgery and with realistic expectation.
* Availability, willingness and sufficient cognitive awareness to comply with examination procedures
* Signed informed consent

Exclusion Criteria:

* Irregular astigmatism
* Age of patient < 50 years
* Regular corneal astigmatism >1.00 dioptres by an automatic keratometer or biometer or >1.25 dioptres if the steep axis of cylinder is between 90° and 120° in one or both eyes
* Difficulty for cooperation (distance from their home, general health condition)
* Acute or chronic disease or illness that would increase risk or confound study results (e.g. diabetes mellitus (with retinopathy), immunocompromised, glaucoma etc…)
* Any ocular comorbidity
* History of ocular trauma or prior ocular surgery including refractive procedures
* Capsule or zonular abnormalities that may affect postoperative centration or tilt of the lens (e.g. pseudoexfoliation syndrome, chronic Uveitis, Marfan's syndrome)
* Pupil abnormalities (non-reactive, tonic pupils, abnormally shaped pupils or pupils that do not dilate under mesopic/scotopic conditions)
* AMD suspicious eyes (determined by OCT)
* Complicated surgery

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2017-10-02 (Actual); Primary Completion 2019-05-21 (Actual); Study Completion 2019-05-21 (Actual)

PRIMARY OUTCOMES:
monocular Uncorrected Distance Visual Acuity (UDVA) under photopic light conditions. | 3 months postoperative
  The primary study end point is to show statistically equal visual acuity outcomes between both study groups. The primary study endpoint parameter is monocular Uncorrected Distance Visual Acuity (UDVA) under photopic light conditions. UDVA is measured with ETDRS charts placed in 4m distance according to ISO 11979-7:2014

SECONDARY OUTCOMES:
Manifested refraction - Sphere | 3 months postoperative
  The spherical part of the manifested refraction is measured by means of a phoropter. The examination is done according to ISO 11979-7:2014.
Manifested refraction - Cylinder | 3 months postoperative
  The cylindrical part of the manifested refraction is measured by means of a phoropter. Amount of cylinder and cylinder axis will be noted. The examination is done according to ISO 11979-7:2014. This data will also be used to calculate the manifested refractive spherical equivalent (MRSE)
Uncorrected Distance Visual Acuity (UDVA) | 3 months postoperative
  UDVA is measured with ETDRS charts placed in 4m distance according to ISO 11979-7:2014. This assessment is done binocularly.
Corrected Distance Visual Acuity (CDVA) | 3 months postoperative
  CDVA is measured with ETDRS charts placed in 4m distance with best aided corrective glasses according to ISO 11979-7:2014. This assessment is done monocularly and binocularly.
Distance Corrected Intermediate Visual Acuity at 80cm (DCIVA) | 3 months postoperative
  DCIVA is measured with Radner reading charts placed in 80cm distance with corrective glasses for far distance according to ISO 11979-7:2014. This assessment is done monocularly and binocularly.
Distance Corrected Intermediate Visual Acuity at 63cm (DCIVA) | 3 months postoperative
  DCIVA is measured with ETDRS charts placed in 63cm distance with corrective glasses for far distance according to ISO 11979-7:2014. This assessment is done monocularly and binocularly.
Distance Corrected Near Visual Acuity at 40cm (DCNVA) | 3 months postoperative
  DCNVA is measured with Radner reading charts placed in 40cm distance with corrective glasses for far distance according to ISO 11979-7:2014. This assessment is done monocularly and binocularly.
Distance Corrected Near Visual Acuity at 25cm (DCNVA) | 3 months postoperative
  DCNVA is measured with Radner reading charts placed in 25cm distance with corrective glasses for far distance according to ISO 11979-7:2014. This assessment is done monocularly and binocularly.
Halometry | 3 months postoperative
  Halometry outcomes, measurement by halos software v1.0
Contrast Sensitivity | 3 months postoperative
  Contrast Sensitivity under photopic and mesopic light conditions using the standardized contrast sensitivity device CSV-1000 (VectorVision)
Aberrometry - SA | 3 months postoperative
  Aberrometry outcomes are measured with a standard aberrometer. In this examination, the following values will be evaluated: Spherical aberration
Aberrometry - HOA | 3 months postoperative
  Aberrometry outcomes are measured with a standard aberrometer. In this examination, the following values will be evaluated: High Order Aberrations
Aberrometry - Tilt | 3 months postoperative
  Aberrometry outcomes are measured with a standard aberrometer. In this examination, the following values will be evaluated: lens tilt
OQAS II - OSI | 3 months postoperative
  Outcomes of OQAS II diagnostic device (Ocular Scatter Index)
OQAS II - MTF | 3 months postoperative
  Outcomes of OQAS II diagnostic device (Modular Transfer Function)
OQAS II - Strehl Ratio | 3 months postoperative
  Outcomes of OQAS II diagnostic device (Strehl Ratio)
questionnaire | 3 months postoperative
  Outcomes measures of a questionnaire to address the general patient satisfaction and possible side effects of the treatment. For this study, the validated and verified questionnaire VFQ-25 (National Eye Institute) will be used. The maximum score for each question is 100. The scoring and evaluation of the questionnaire will be done according to the official guidelines and manual provided by National Eye Institute

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Poyales Galan, MD, Principal Investigator — Innova Ocular IOA Madrid
Locations (1):
- Innova Ocular IOA Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No